CLINICAL TRIAL: NCT04455529
Title: A Research of Current Situation of Natural History, Diagnosis and Treatment in Inpatients With Embolism Stroke of Unknown Cause (ESUS)
Brief Title: Current Situation of Natural History, Diagnosis and Treatment in Inpatients With Embolism Stroke of Unknown Cause (ESUS)
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PUTH2016144
Record Dates: First submitted 2020-06-28; First posted 2020-07-02 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-06

CONDITIONS: Embolic Stroke of Undetermined Source

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ESUS: Embolic stroke of undetermined source (ESUS) designates patients with nonlacunar cryptogenic ischemic strokes in whom embolism is the likely stroke mechanism.
  Interventions: Other: ESUS

INTERVENTIONS:
Other: ESUS — Embolic stroke of undetermined source (ESUS) designates patients with nonlacunar cryptogenic ischemic strokes in whom embolism is the likely stroke mechanism.

SUMMARY:
Evaluate the epidemiological characteristics, risk factors, clinical characteristics in patients with ESUS and their medication compliance and relapse within 1 year.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the epidemiological characteristics, risk factors (such as hypertension, diabetes, hyperlipidemia, coronary heart disease, history of previous stroke, smoking, and alcohol consumption), clinical characteristics in patients with ESUS and their medication compliance and relapse within 1 year.

ELIGIBILITY:
Inclusion Criteria:

- Patients diagnosed with acute cerebral infarction and treated in Peking University Third Hospital Neurology Department from January 2010 to June 2016.

Exclusion Criteria:

* Lacunar infarction
* Aortic atherosclerotic cerebral infarction
* Clear cardiogenic cerebral infarction
* Other related system diseases (arteritis, vascular dissection, migraine and vasospasm, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We recruited consecutive patients with Embolism Stroke of Unknown Cause.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
Medication adherence | 1 year after recruitment
  Medication adherence usually refers to whether patients take their medications as prescribed (eg, twice daily), as well as whether they continue to take a prescribed medication. The Morisky scale, a validated, 4-item self-reported adherence measure that has been shown to be predictive of adherence to cardiovascular medications and blood pressure control. If a patient scores higher on the scale, they are evaluated as more adherent. If they score lower on the scale, they are presumed to be struggling with nonadherence.
Recurrence rate | 1 year after recruitment
  Recurrence rate of stroke

CONTACTS AND LOCATIONS:
Overall Officials: Dongsheng Fan, MD.PHD, Principal Investigator — Peking University Third Hospital

IPD SHARING:
Plan to Share IPD: No